CLINICAL TRIAL: NCT00800176
Title: A Multi-center, Double-blind, Randomized, Parallel Group, Placebo-controlled 12-week Study to Investigate Glycemic Parameters of Efficacy, Safety/ Tolerability and Pharmacokinetics of Five Dose Levels of RO4998452 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Dose-Finding Study of RO4998452 in Patients With Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC21587; 2008-001249-24
Record Dates: First submitted 2008-12-01; First posted 2008-12-02 (Estimated); Results first posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Placebo (Placebo Comparator): During the single-blind run-in period, two placebo capsules were taken in the morning approximately 15 minutes prior to breakfast.
  During the 12-week double-blind treatment period, two placebo capsules were taken in the morning approximately 15 minutes prior to breakfast, except on the days of the meal tolerance test.
  Interventions: Drug: Placebo
- RO4998452 10mg (Experimental): During the single-blind run-in period, two placebo capsules were taken in the morning approximately 15 minutes prior to breakfast. During the 12-week double-blind treatment period, two capsules were taken in the morning approximately 15 minutes prior to breakfast, except on the days of the meal tolerance test. The two capsules combined contained 10 mg of RO4998452.
  Interventions: Drug: RO4998452
- RO4998452 2.5mg (Experimental): During the single-blind run-in period, two placebo capsules were taken in the morning approximately 15 minutes prior to breakfast. During the 12-week double-blind treatment period, two capsules were taken in the morning approximately 15 minutes prior to breakfast, except on the days of the meal tolerance test. The two capsules combined contained 2.5 mg of RO4998452.
  Interventions: Drug: RO4998452
- RO4998452 20mg (Experimental): During the single-blind run-in period, two placebo capsules were taken in the morning approximately 15 minutes prior to breakfast. During the 12-week double-blind treatment period, two capsules were taken in the morning approximately 15 minutes prior to breakfast, except on the days of the meal tolerance test. The two capsules combined contained 20 mg of RO4998452.
  Interventions: Drug: RO4998452
- RO4998452 40mg (Experimental): During the single-blind run-in period, two placebo capsules were taken in the morning approximately 15 minutes prior to breakfast. During the 12-week double-blind treatment period, two capsules were taken in the morning approximately 15 minutes prior to breakfast, except on the days of the meal tolerance test. The two capsules combined contained 40 mg of RO4998452.
  Interventions: Drug: RO4998452
- RO4998452 5mg (Experimental): During the single-blind run-in period, two placebo capsules were taken in the morning approximately 15 minutes prior to breakfast. During the 12-week double-blind treatment period, two capsules were taken in the morning approximately 15 minutes prior to breakfast, except on the days of the meal tolerance test. The two capsules combined contained 5 mg of RO4998452.
  Interventions: Drug: RO4998452

INTERVENTIONS:
Drug: Placebo — po daily for 12 weeks
  Arms: Placebo
Drug: RO4998452 — 2.5mg po daily for 12 weeks
  Arms: RO4998452 2.5mg
Drug: RO4998452 — 5mg po daily for 12 weeks
  Arms: RO4998452 5mg
Drug: RO4998452 — 10mg po daily for 12 weeks
  Arms: RO4998452 10mg
Drug: RO4998452 — 20mg po daily for 12 weeks
  Arms: RO4998452 20mg
Drug: RO4998452 — 40mg po daily for 12 weeks
  Arms: RO4998452 40mg

SUMMARY:
This 6 arm study will evaluate the efficacy, safety and pharmacokinetics of 5 doses of RO4998452 compared to placebo in patients with type 2 diabetes mellitus. Patients will be randomized to one of 6 groups to receive RO4998452 at doses of 2.5mg, 5mg, 10mg, 20mg or 40mg po daily, or placebo daily. Patients pre-treated with stable metformin will continue to take their usual dose of metformin throughout the study.The anticipated time on study treatment is <=3 months

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes, diagnosed for >=3 months;
* either treated with diet, exercise and stable metformin, or with diet and exercise alone.

Exclusion Criteria:

* type 1 diabetes mellitus;
* currently or within 2 months prior to screening treated with an oral or injectable anti-diabetic agent except stable doses of metformin;
* currently or within 6 months prior to screening treated with any PPARgamma agonist;
* uncontrolled hypertension;
* significant pre-diagnosed diabetic complications requiring treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2009-01-22 (Actual); Primary Completion 2009-10-28 (Actual); Study Completion 2009-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (53):
- United States (11):
  - Phoenix, Arizona
  - Los Angeles, California
  - Palm Springs, California
  - Bradenton, Florida
  - Jacksonville, Florida
  - Atlanta, Georgia
  - Hayden Lake, Idaho
  - Rochester, New York
  - Greensboro, North Carolina
  - Midland, Texas
  - Richmond, Virginia
- Australia (2):
  - Adelaide
  - St Leonards
- Brazil (3):
  - Fortaleza
  - Goiânia
  - São Paulo
- Canada (4):
  - Vancouver, British Columbia
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- Germany (5):
  - Berlin
  - Falkensee
  - Lübeck
  - Mainz
  - Neuss
- Hong Kong, Hong Kong
- Japan (6):
  - Fukuoka
  - Ibaraki
  - Kanagawa
  - Osaka
  - Saitama
  - Tokyo
- Latvia (4):
  - Jelgava
  - Riga
  - Talsi
  - Valmiera
- Mexico (3):
  - Chihuahua City
  - Guadalajara
  - Mexico City
- Romania (4):
  - Alba Iulia
  - Brasov
  - Bucharest
  - Târgu Mureş
- Russia (7):
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - S.petersburg
  - Saint Petersburg
  - Saratov
  - Yaroslavl
- Spain (3):
  - Alzira
  - Lleida
  - Seville

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening period: Week 6 to 5 prior to randomization
Pre-assignment Details: As soon as the results of the screening tests were available, eligible patients could start the 4-week placebo run-in period (visit week -4). A diet and exercise plan was discussed based on the recommendations of the investigator. This plan was not to be changed during the study
Groups:
- RO4998452 10 mg: During the single-blind run-in period, two placebo capsules were taken in the morning approximately 15 minutes prior to breakfast. During the 12-week double-blind treatment period, two capsules were taken in the morning approximately 15 minutes prior to breakfast, except on the days of the meal tolerance test. The two capsules combined contained 10 mg of RO4998452.
Period: Overall Study
Arm/Group | Placebo | RO4998452 2.5mg | RO4998452 5mg | RO4998452 10 mg | RO4998452 20mg | RO4998452 40mg
Started | 66 | 66 | 65 | 66 | 64 | 67
Completed | 57 | 60 | 65 | 62 | 60 | 62
Not Completed | 9 | 6 | 0 | 4 | 4 | 5
Not completed — Adverse Event | 2 | 1 | 0 | 2 | 1 | 1
Not completed — Refused treatment | 3 | 2 | 0 | 0 | 1 | 4
Not completed — Failure to return | 3 | 3 | 0 | 2 | 0 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The safety population was used for baseline characteristics. The safety population consisted of all patients randomized and received at least one dose of double-blind study medication (DBSM). If patient received incorrect dose of DBSM throughout study, patient was analyzed according to dose actually received. If patient received an incorrect dose of DBSM for only a portion of study, patient was analyzed according to dose patient was randomized to.
Groups:
- RO4998452 2.5 mg: During the single-blind run-in period, two placebo capsules were taken in the morning approximately 15 minutes prior to breakfast. During the 12-week double-blind treatment period, two capsules were taken in the morning approximately 15 minutes prior to breakfast, except on the days of the meal tolerance test. The two capsules combined contained 2.5 mg of RO4998452.
- Total: Total of all reporting groups
Arm/Group | Placebo | RO4998452 2.5 mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg | Total
Number analyzed (Participants) | 66 | 66 | 65 | 66 | 64 | 67 | 394
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.9 (11.12) | 53.3 (10.86) | 54.8 (10.53) | 54.5 (10.7) | 56.3 (9.79) | 57.5 (9.31) | 55.1 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 34 | 32 | 21 | 36 | 185
  Male | 36 | 34 | 31 | 34 | 43 | 31 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 46 | 41 | 40 | 45 | 39 | 253
  Not Hispanic or Latino | 24 | 20 | 24 | 26 | 19 | 28 | 141
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 18 | 14 | 14 | 15 | 13 | 19 | 93
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2 | 2 | 0 | 6
  White | 42 | 46 | 41 | 40 | 45 | 39 | 253
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 6 | 9 | 9 | 4 | 9 | 42
Race/Ethnicity, Customized [Number; unit: Participants]
  Ex-Japan | 54 | 55 | 53 | 54 | 53 | 54 | 323
  Japan | 12 | 11 | 12 | 12 | 11 | 13 | 71

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in HbA1c
Time Frame: Baseline, Week 4, Week 8 and Week 12
Population: Full analysis set included all patients who were randomized, received at least one dose of study medication, and had an evaluable baseline and at least one evaluable post baseline measurement of HbA1c. If patient's HbA1c value at baseline visit was missing, latest screening HbA1c value was used as baseline. If patient received an incorrect dose of study medication at any time during study, patient was analyzed according to dose patient was randomized to, not dose patient received.
Measure: Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo | RO4998452 2.5 mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg
Number analyzed (Participants) | 65 | 64 | 65 | 66 | 64 | 66
Percentage
  Baseline | 7.872 [7.695 to 8.049] | 7.939 [7.829 to 8.118] | 8.006 [7.823 to 8.183] | 7.998 [7.823 to 8.174] | 7.919 [7.740 to 8.097] | 7.933 [7.758 to 8.109]
  Week 4: number analyzed (Participants) | 63 | 64 | 65 | 65 | 64 | 66
  Week 4 | -0.238 [-0.341 to -0.135] | -0.394 [-0.497 to -0.291] | -0.460 [-0.561 to -0.358] | -0.539 [-0.641 to -0.437] | -0.516 [-0.619 to -0.413] | -0.564 [-0.664 to -0.464]
  Week 8 | -0.280 [-0.405 to -0.155] | -0.468 [-0.594 to -0.342] | -0.611 [-0.736 to -0.486] | -0.694 [-0.840 to -0.549] | -0.768 [-0.916 to -0.620] | -0.832 [-0.976 to -0.688]
  Week 12 | -0.269 [-0.415 to -0.123] | -0.440 [-0.588 to -0.293] | -0.617 [-0.763 to -0.471] | -0.694 [-0.840 to -0.549] | -0.768 [-0.916 to -0.620] | -0.832 [-0.976 to -0.688]

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (mmol/L)
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | RO4998452 2.5 mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg
Number analyzed (Participants) | 65 | 64 | 65 | 66 | 64 | 66
mmol/L
  Baseline | 8.738 [8.312 to 9.164] | 8.917 [8.488 to 9.347] | 8.695 [8.269 to 9.121] | 8.824 [8.401 to 9.247] | 8.741 [8.311 to 9.170] | 8.992 [8.570 to 9.415]
  Last Visit: Change from Baseline: number analyzed (Participants) | 65 | 64 | 65 | 65 | 63 | 65
  Last Visit: Change from Baseline | -0.502 [-0.854 to -0.149] | -0.021 [-0.376 to 0.335] | -0.641 [-0.993 to -0.288] | -1.042 [-1.395 to -0.690] | -0.935 [-1.294 to -0.577] | -1.422 [-1.771 to -1.073]

3. Secondary Outcome: Change From Baseline in Mean Daily Glucose Concentration (mmol/L)
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | RO4998452 2.5 mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg
Number analyzed (Participants) | 65 | 64 | 63 | 66 | 64 | 66
mmol/L
  Change from Baseline | 9.655 [9.236 to 10.075] | 9.546 [9.123 to 9.968] | 9.750 [9.324 to 10.176] | 9.843 [9.427 to 10.259] | 9.614 [9.192 to 10.037] | 9.648 [9.232 to 10.064]
  Last Visit: Absolute Change from Baseline: number analyzed (Participants) | 64 | 64 | 63 | 65 | 63 | 65
  Last Visit: Absolute Change from Baseline | -0.278 [-0.599 to 0.043] | -0.556 [-0.878 to -0.233] | -0.800 [-1.123 to -0.477] | -1.055 [-1.375 to -0.734] | -0.882 [-1.207 to -0.558] | -1.298 [-1.615 to -0.981]

4. Secondary Outcome: Change From Baseline in Fructosamine Concentration (μmol/L)
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: μmol/L
Arm/Group | Placebo | RO4998452 2.5 mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg
Number analyzed (Participants) | 65 | 64 | 65 | 66 | 64 | 66
μmol/L
  Baseline | 293.292 [283.047 to 303.538] | 294.891 [284.566 to 305.216] | 292.600 [282.355 to 302.845] | 290.970 [280.802 to 301.137] | 292.672 [282.347 to 302.997] | 305.015 [294.848 to 315.182]
  Last Visit: Absolute Change from Baseline: number analyzed (Participants) | 55 | 58 | 65 | 61 | 59 | 59
  Last Visit: Absolute Change from Baseline | -0.368 [-8.417 to 7.680] | -11.202 [-19.092 to -3.312] | -12.992 [-20.491 to -5.493] | -16.712 [-24.411 to -9.013] | -18.758 [-26.583 to -10.934] | -20.619 [-28.446 to -12.792]

5. Secondary Outcome: Change From Baseline in Meal Tolerance Test: 0-3h Mean Glucose Concentration (mmol/L)
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | RO4998452 2.5 mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg
Number analyzed (Participants) | 63 | 63 | 65 | 66 | 63 | 65
mmol/L
  Baseline | 11.663 [11.119 to 12.207] | 11.661 [11.116 to 12.205] | 11.689 [11.153 to 12.225] | 11.432 [10.900 to 11.963] | 11.643 [11.099 to 12.187] | 12.032 [11.496 to 12.568]
  Last Visit: Absolute Change from Baseline: number analyzed (Participants) | 54 | 56 | 61 | 59 | 59 | 57
  Last Visit: Absolute Change from Baseline | -0.655 [-1.053 to -0.257] | -1.692 [-2.083 to -1.301] | -2.146 [-2.522 to -1.769] | -2.347 [-2.731 to -1.964] | -2.443 [-2.827 to -2.059] | -2.884 [-3.268 to -2.501]

6. Secondary Outcome: Change From Baseline in Meal Tolerance Test: 0-3h Mean Insulin Concentration (mmol/L)
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | RO4998452 2.5 mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg
Number analyzed (Participants) | 59 | 61 | 62 | 64 | 61 | 63
mmol/L
  Baseline | 201.243 [169.516 to 232.970] | 202.269 [171.066 to 233.471] | 207.255 [176.305 to 238.204] | 223.964 [193.501 to 254.426] | 219.396 [188.194 to 250.599] | 189.286 [158.583 to 219.989]
  Last Visit: Absolute Change from Baseline: number analyzed (Participants) | 50 | 52 | 58 | 54 | 55 | 54
  Last Visit: Absolute Change from Baseline | -8.909 [-26.748 to 8.929] | -46.108 [-63.662 to -28.553] | -39.409 [-56.095 to -22.723] | -68.881 [-86.116 to -51.647] | -67.373 [-84.466 to -50.281] | -58.053 [-75.228 to -40.878]

7. Secondary Outcome: Change From Baseline in Meal Tolerance Test: 0-3h Urinary Glucose Excretion (mmol/L)
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | RO4998452 2.5 mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg
Number analyzed (Participants) | 63 | 64 | 63 | 65 | 62 | 66
mmol/L
  Baseline | 6.607 [2.098 to 11.116] | 8.472 [3.999 to 12.946] | 6.841 [2.332 to 11.350] | 11.659 [7.220 to 16.098] | 14.039 [9.494 to 18.585] | 10.395 [5.990 to 14.801]
  Last Visit: Absolute Change from Baseline: number analyzed (Participants) | 52 | 57 | 60 | 59 | 57 | 57
  Last Visit: Absolute Change from Baseline | -1.282 [-13.644 to 11.079] | 43.369 [31.519 to 55.219] | 52.396 [40.818 to 63.975] | 68.634 [56.957 to 80.311] | 62.610 [50.694 to 74.527] | 59.294 [47.550 to 71.038]

8. Secondary Outcome: Change From Baseline in Body Weight (kg)
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Placebo | RO4998452 2.5 mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg
Number analyzed (Participants) | 65 | 64 | 65 | 66 | 64 | 66
kg
  Baseline | 83.965 [79.691 to 88.238] | 85.455 [81.148 to 89.762] | 82.149 [77.876 to 86.423] | 83.411 [79.169 to 87.652] | 84.914 [80.607 to 89.221] | 81.568 [77.327 to 85.809]
  Last Visit: Absolute Change from Baseline | -0.741 [-1.218 to -0.265] | -1.564 [-2.044 to -1.083] | -1.853 [-2.332 to -1.375] | -2.235 [-2.711 to -1.759] | -2.551 [-3.032 to -2.070] | -2.824 [-3.297 to -2.351]

9. Secondary Outcome: Percentage of Participants Treated to Target HbA1c < 7%
Time Frame: Baseline up to 12 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo | RO4998452 2.5 mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg
Number analyzed (Participants) | 65 | 64 | 65 | 66 | 64 | 66
Percentage | 13.8 [6.5 to 24.7] | 17.2 [8.9 to 28.7] | 23.1 [13.5 to 35.2] | 24.2 [14.5 to 36.4] | 34.4 [22.9 to 47.3] | 40.9 [29.0 to 53.7]

10. Secondary Outcome: Percentage of Participants Treated to Target HbA1c < 6.5%
Time Frame: Baseline up to 12 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Placebo | RO4998452 2.5 mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg
Number analyzed (Participants) | 65 | 64 | 65 | 66 | 64 | 66
Percentage | 3.1 [0.4 to 10.7] | 6.3 [1.7 to 15.2] | 9.2 [3.5 to 19.0] | 6.1 [1.7 to 14.8] | 10.9 [4.5 to 21.2] | 16.7 [8.6 to 27.9]

11. Secondary Outcome: Percentage of Participants With at Least One Adverse Event
Time Frame: Baseline up to 12 weeks
Population: The safety population consisted of all patients randomized and received at least one dose of double-blind study medication (DBSM). If patient received incorrect dose of DBSM throughout study, patient was analyzed according to dose actually received. If patient received an incorrect dose of DBSM for only a portion of study, patient was analyzed according to dose patient was randomized to.
Measure: Number; unit: Percentage
Arm/Group | Placebo | RO4998452 2.5 mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg
Number analyzed (Participants) | 66 | 66 | 65 | 66 | 64 | 67
Percentage | 37.9 | 36.4 | 46.2 | 37.9 | 35.9 | 46.3

ADVERSE EVENTS:
Time Frame: Baseline up to 8 months
Description: The safety population consisted of all patients randomized and received at least one dose of double-blind study medication (DBSM). If patient received incorrect dose of DBSM throughout study, patient was analyzed according to dose actually received. If patient received an incorrect dose of DBSM for only a portion of study, patient was analyzed according to dose patient was randomized to.
Arm/Group | Placebo | RO4998452 2.5mg | RO4998452 5mg | RO4998452 10mg | RO4998452 20mg | RO4998452 40mg
Serious Adverse Events (participants affected / at risk) | 1/66 | 2/66 | 0/65 | 0/66 | 0/64 | 1/67
Other Adverse Events (participants affected / at risk) | 25/66 | 24/66 | 30/65 | 25/66 | 23/64 | 31/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=66) | RO4998452 2.5mg (N=66) | RO4998452 5mg (N=65) | RO4998452 10mg (N=66) | RO4998452 20mg (N=64) | RO4998452 40mg (N=67)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=66) | RO4998452 2.5mg (N=66) | RO4998452 5mg (N=65) | RO4998452 10mg (N=66) | RO4998452 20mg (N=64) | RO4998452 40mg (N=67)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
PHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CERVICITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DENGUE FEVER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FURUNCLE (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GENITAL INFECTION FUNGAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GENITOURINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTITIS EXTERNA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TINEA PEDIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
GINGIVAL PAIN (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTRA-ABDOMINAL HAEMATOMA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SALIVA ALTERED (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
DIZZINESS (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
DIABETIC NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUS HEADACHE (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
APHONIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BURNING SENSATION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FACIAL PALSY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERSOMNIA (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCIATICA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INTERVERTEBRAL DISC (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCLE CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INCREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
POLYDIPSIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD FIBRINOGEN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM T WAVE ABNORMAL (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLOOD UREA INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM REPOLARISATION ABNORMALITY (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ELECTROCARDIOGRAM T WAVE BIPHASIC (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HELICOBACTER PYLORI IDENTIFICATION TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LYMPH NODE PALPABLE (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINE OUTPUT INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POLLAKIURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MICTURITION URGENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POLYURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RENAL IMPAIRMENT (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PALPITATIONS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HUNGER (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
THIRST (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VESSEL PUNCTURE SITE HAEMATOMA (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
EPICONDYLITIS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
JOINT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERIORBITAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THERMAL BURN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ANXIETY (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
AGITATION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LIBIDO DECREASED (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOSS OF LIBIDO (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIABETIC RETINOPATHY (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GLAUCOMA (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OCULAR DISCOMFORT (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OCULAR HYPERAEMIA (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISUAL ACUITY REDUCED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RASH PRURITIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SKIN EROSION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MENORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
METRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRURITUS GENITAL (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HOT FLUSH (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (11) | 0 (0)
PHIMOSIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TYPE II HYPERLIPIDAEMIA (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TYPE IV HYPERLIPIDAEMIA (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DENTAL IMPLANTATION (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOOTH EXTRACTION (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.